CLINICAL TRIAL: NCT04547556
Title: ADEQUATE Advanced Diagnostics for Enhanced QUality of Antibiotic Prescription in Respiratory Tract Infections in Emergency Rooms
Brief Title: ADEQUATE Advanced Diagnostics for Enhanced Quality of Antibiotic Prescription
Acronym: ADEQUATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment in the context of the pandemic.
Sponsor: UMC Utrecht (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Dr. Cristina Prat, Sponsor Central Principal Investigator: Dr. C. Prat, MD, PhD, Microbiologist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WP4b - adults
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Diagnostic intervention
  Interventions: Diagnostic Test: BioFire
- Standard of Care (No Intervention): Standard of care testing

INTERVENTIONS:
Diagnostic Test: BioFire — A molecular rapid syndromic testing platform, using the following panels:
  * BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus)
  * BioFire FilmArray Pneumonia Panel plus (PP)
  Arms: Intervention

SUMMARY:
To assess the impact of rapid diagnostic testing of patients with Acute Respiratory Tract Infection (ARTI) at the emergency department, on (1) hospital admission rates and (2) antimicrobial prescriptions (days of treatment) and (3) the non-inferiority in terms of clinical outcome. Geographical and seasonal variation will be assessed on a real time basis including pathogens of public health interest. The impact will be stratified within age groups and risk factors in order to determine the long-term clinical, public health and economic determinants for the integration of diagnostics in a global and sustainable perspective.

DETAILED DESCRIPTION:
Objective: To assess the impact of rapid diagnostic testing of patients with Acute Respiratory Tract Infection (ARTI) at the emergency department, on (1) hospital admission rates and (2) antibiotic prescriptions (days of treatment) and (3) the non-inferiority in terms of clinical outcome. Geographical and seasonal variation will be assessed on a real time basis including pathogens of public health interest. The impact will be stratified within age groups and risk factors in order to determine the long-term clinical, public health and economic determinants for the integration of diagnostics in a global and sustainable perspective.

Study design: Prospective, multi-center, individually randomised, controlled trial.

Study population: Adults (≥18 years old) consulting in selected participating sites with CA-ARTI.

Study Intervention: The diagnostic intervention is rapid syndromic testing with:

* BioFire FilmArray Pneumonia Panel plus (PP): Sputum (and/or ETA or BAL sample)
* BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus): Nasopharyngeal swab

Main study parameters/endpoints:

* Days alive out of hospital (superiority endpoint), within 14 days
* Days on Therapy (DOT) with antibiotics (superiority endpoint), within 14 days
* Adverse outcome (non-inferiority safety endpoint)

  * For initially non-admitted patients: any admission or death within 30 days
  * For initially hospitalised patients: i) any readmission, ii) ICU admission ≥ 24 hours after hospitalisation, or iii) death within 30 days Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in the study involves collection of data that can be obtained from medical charts and follow up questionnaires and interviews. Respiratory samples (e.g. nasopharyngeal swab, sputum) will be obtained as standard of care and diagnostic intervention (Biofire FilmArray) will be used only for participants randomised to the intervention,Based on the results of diagnostic testing (BioFire FilmArray) antibiotics may be withheld when deemed unnecessary, or a different antibiotic class may be selected when certain bacterial pathogens are detected. The risks and benefits of management decisions, complemented with adequate training, are subject to the current investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old) presenting to the Emergency Room with an acute illness (present for 14 days or less) with cough, and with at least 1 other lower respiratory tract symptom or clinical sign at physical examination:

   * Sputum production,
   * Breathlessness,
   * Chest discomfort or chest pain,
   * Wheeze,
   * Crackles,
   * Self-reported dystermia or documented fever;
   * Documented hypoxemia (adjusting definition for chronic oxygen therapy users, method of measurement) and no alternative explanation (infection, such as sinusitis; other, such as asthma).

     2. Managing medical team considers:
     1. to treat patient with antibiotics and/or to hospitalize patient

        AND
     2. that the rapid syndromic diagnostic test result can be awaited up to a maximum of 4 hours before the decision to discharge the patient or to initiate antibiotic therapy.

Exclusion Criteria:

1. Development of ARTI more than 48 hours after hospital admission (hospital acquired);
2. Patients with cystic fibrosis;
3. Less than 14 days since the last episode of respiratory tract infection;
4. Pregnancy (confirmed by pregnancy test) and breastfeeding;
5. Any clinically significant abnormality identified at the time of screening that in the judgment of the Investigator would preclude safe completion of the study or constrain endpoints assessment such as major systemic diseases or patients with short life expectancy;
6. Inability to obtain informed consent from a competent patient.

   Based on standard of care microbiological diagnosis and thoracic imaging (when indicated):
7. Radiologically confirmed acute lobar pneumonia;
8. Known or suspected Pneumocystis jirovecii pneumonia or active tuberculosis;
9. Alternative noninfectious diagnosis that explains clinical symptoms (pulmonary embolism, alveolar hemorrhage, acute heart failure, lung cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, MD, Principal Investigator — UMC Utrecht
Locations (4):
- University Hospital Gent, Ghent, Belgium
- University Hospital Pecs, Pécs, Hungary
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - General Hospital Kragujevac, Kragujevac

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of care diagnostics
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 92 | 93
Completed | 92 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Standard of care diagnostic testing
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 92 | 93 | 185
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.5 [58 to 75] | 67 [48 to 78] | 67 [53 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 91
  Male | 46 | 48 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Serbia | 88 | 91 | 179
  Belgium | 3 | 2 | 5
  Hungary | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Days Alive Out of Hospital (Superiority Endpoint)
Description: Days alive out of hospital (superiority endpoint), within 14 days after study enrolment
Time Frame: Day 1 - Day 14
Population: Days alive out of hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
days | 10.7 (5.3) | 9.7 (5.9)

2. Primary Outcome: Days on Therapy (DOT) With Antibiotics (Superiority Endpoint)
Description: Days on Therapy (DOT) with antibiotics (superiority endpoint), within 14 days after study enrolment
Time Frame: Day 1 - Day 14
Population: Number of antibiotic treatment days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
days | 6.7 (4.6) | 7 (4.7)

3. Primary Outcome: Adverse Outcome (Non-inferiority Safety Endpoint)
Description: * For initially non-admitted patients: any admission or death
  * For initially hospitalized patients: any readmission, ICU admission >= 24 hours after hospitalization, or death
Time Frame: Day 1 - Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
Participants | 9 | 18

4. Secondary Outcome: Direct Costs and Indirect Costs Within 30 Days After Enrolment.
Description: * Cost of healthcare within 30 days after enrolment, including hospital and ICU days, utilisation of non-hospital services and cost of anti-infective and concomitant medication
  * Cost of workdays lost within 30 days, including days for childcare
Time Frame: Day 1 - Day 30
Population: This outcome will not be analysed since direct costs and indirect costs could not be properly collected. Cost effective algorithms might change with factors as the disease incidence changes, performance of other diagnostic tests or its combination. As these other factors are also dependent on country and vary over time, the data as collected in the trial is insufficient to reliably report on cost-effectiveness in general
Groups:
- Intervention: Diagnostic intervention
  BioFire: A molecular rapid syndromic testing platform, using the following panels:
  * BioFire FilmArray Respiratory Panel 2.1 plus (RP2.1plus)
  * BioFire FilmArray Pneumonia Panel plus (PP)
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Microbiological Results Obtained as Standard of Care and With the Diagnostic Intervention
Description: Proportion of participants with an identified respiratory pathogen in both study groups on randomisation day samples.
  Data refers to the number of participants so in case more than one microorganism is detected in the same sample (co-detection) or same result in more than one sample, it is still counted as one participant.
Time Frame: Day 1
Population: Data collected includes: sample type (upper and lower respiratory tract samples for diagnostic intervention but also blood cultures and urinary antigen tests for standard of care if applicable), type of diagnostic test, specific results. Data is also collected regarding the time elapsed until the results were received. Results are final for this trial and later on will be compared with pediatric trial results NCT04781530.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
Participants | 58 | 31

6. Secondary Outcome: Empirical Antibiotics Based on Antimicrobial Agent Categories
Description: Proportion of participants on non-first-line anti-infective regimens (as defined by local guidelines).
  For this report, results are defined as non first-line if the choice includes a third or fourth generation cephalosporin or a carbapenem but analysis needs to be adjusted to baseline risk factors, comorbidities, local guidelines and time to de escalation.
Time Frame: Day 1 - Day 14
Population: Final analysis needs to integrate data from both the adult and the pediatric protocol and to adjust to local guidelines per country as well as risk factors and comorbidities. Data collected includes: antibiotics, antivirals and antifungals recording if initial, switch or addition to ongoing therapy as well as route of administration, dosing interval and start and stop date.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
Participants | 30 | 33

7. Secondary Outcome: Antibiotic Type Switches and De-escalation Based on Antimicrobial Agent Categories
Description: For this report is presented the number of patients where the antimicrobial was switched to narrower spectrum.
Time Frame: Day 1 - Day 14
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 92 | 93
Participants | 11 | 15

8. Secondary Outcome: Detection of Antimicrobial Resistance (Carriage or Infection) Related to the Diagnostic Intervention Results Compared to Standard of Care and Impact on Antimicrobial Stewardship Guidelines and Prevention of Hospital Acquired Infections.
Description: Proportion of hospitalised participants with detection of cephalosporin-, carbapenem- or chinolone-resistant Enterobacteriaceae on any standard of care samples >7 days after randomisation comparing diagnostic intervention arm and standard of care arm.
Time Frame: >7 days after randomisation
Population: Hospitalised participants. Samples obtained as standard of care during hospital stay. Detection of multidrug resistant microorganism was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 27 | 32
Participants | 0 | 0

9. Secondary Outcome: Impact on Decisions Regarding Isolation Measures Related to Test Result.
Description: Hours in individual or cohort isolation in hospitalised participants comparing the 2 groups
Time Frame: Day 1 - Day 30
Population: Hospitalised participants. Data collected includes start and stop date of individual or cohort isolation. Isolation measures in the current cohort were related to SARS-CoV-2 infection and not to the detection of multidrug resistant bacteria.
Measure: Median (Standard Deviation); unit: hours in isolation
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 27 | 32
hours in isolation | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent through study completion (day-30 for the main study or 6 months for the extension study).
Description: Standard definitions of adverse events and device related events.
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 5/92 | 11/93
Serious Adverse Events (participants affected / at risk) | 5/92 | 14/93
Other Adverse Events (participants affected / at risk) | 0/92 | 3/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=92) | Standard of Care (N=93)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4) | 10 (10)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=92) | Standard of Care (N=93)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID 19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The calculated sample size for the trial NCT04547556, which is the adult arm of the ADEQUATE trial could not be achieved and study was terminated due to poor enrolment. Outcome measures that could be calculated are provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT04547556/Prot_SAP_000.pdf